CLINICAL TRIAL: NCT00007592
Title: VA HYPERTENSION SCREENING AND TREATMENT PROGRAM (PILOT STUDY)
Brief Title: Hypertension Screening and Treatment Program
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: 324
Record Dates: First submitted 2000-12-29; First posted 2001-01-01 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2003-02

CONDITIONS: Hypertension
Keywords: Hypertension; national data base on the treatment of hypertension; cost of different antihypertensive regimens
MeSH Terms: conditions — Hypertension | interventions — Chlorthalidone; Furosemide

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Drug: Chlorthalidone
Drug: Furosemide

SUMMARY:
Hypertension is one of the most common medical problems in the United States and in the VA health care system. It has been well-documented that hypertension can be effectively treated. However, there remain important unresolved clinical questions in the area of antihypertensive treatment. For example, how much is mortality affected by visit compliance, blood pressure control and type of antihypertensive agent? Or, are some regimens associated with more morbidity than others? Or, are there inexpensive regimens that are as effective as more expensive regimens? The amount of data that is available from this demonstration project (currently 6,100 patients) will help address these questions. The answers to these questions should result in better care for veterans with hypertension.

DETAILED DESCRIPTION:
Primary Hypothesis: A variety of clinical questions of major importance can be addressed using clinical data routinely obtained in the VA Hypertension Screening and Treatment Program. For example, treatment of mild hypertension reduces the risk of strokes and heart attacks.

Secondary Hypothesis: Target organ damage occurs despite blood pressure control.

Intervention: Chlorthalidone, furosemide, hydrochlorothiazide, metolazone, indapamide, amiloride, spironolactone, triamterene, atenolol, metoprolol, nadolol, pindolol, propranolol, timolol, acebutolol, penbutolol, clonidine, guanethidine, methydopa, prazosin, guanadrel, labetalol, reserpine, guanfacine, hydralazine, minoxidil, captopril, enalapril, lisinopril, diltiazem, nifedipine, verapamil, nicardipine, dyazide, maxzide, pargyline, terazosin, other anti-hypertensives.

Primary Outcomes: Blood Pressure and Target Organ Damage

Study Abstract: Hypertension is one of the most common medical problems in the United States and in the VA health care system. It has been well-documented that hypertension can be effectively treated. However, there remain important unresolved clinical questions in the area of antihypertensive treatment. For example, how much is mortality affected by visit compliance, blood pressure control and type of antihypertensive agent? Or, are some regimens associated with more morbidity than others? Or, are there inexpensive regimens that are as effective as more expensive regimens? The amount of data that is available from this demonstration project (currently 6,100 patients) will help address these questions. The answers to these questions should result in better care for veterans with hypertension.

This demonstration project provides for central collection of a standard set of clinical data for patients at some of the Hypertension Screening and Treatment Program clinics, thereby setting up a national data base on the treatment of hypertension. The primary objective of this project is to demonstrate the value of establishing this type of database. The database is being used to estimate the average annual cost of different antihypertensive regimens, to determine the cost-efficacy of different therapies and the least expensive effective therapy and to address some major unanswered clinical questions that require large populations and long-term patient care data. There are currently 13 medical centers participating.

ELIGIBILITY:
Patients at Hypertension Screening and Treatment Program clinics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1989-06

CONTACTS AND LOCATIONS:
Locations (12):
- United States (11):
  - Vamc - Sepulveda, Sepulveda, California
  - Vamc - Washington, Dc, Washington D.C., District of Columbia
  - Vamc - Miami, Miami, Florida
  - Vamc - Indianapolis, Indianapolis, Indiana
  - Vamc - Iowa City, Iowa City, Iowa
  - Vamc - Jackson, Jackson, Mississippi
  - Vamc - Dayton, Dayton, Ohio
  - Vamc - Philadelphia, Philadelphia, Pennsylvania
  - Vamc - Pittsburgh, Pittsburgh, Pennsylvania
  - Vamc - Memphis, Memphis, Tennessee
  - Vamc - Richmond, Richmond, Virginia
- Vamc - San Juan, Pr, San Juan, Puerto Rico